CLINICAL TRIAL: NCT06662539
Title: A Randomized, Double-blind, Phase 2, Dose-finding Trial of Once Weekly Petrelintide Compared With Placebo in Participants With Obesity or Overweight With Weight Related Comorbidities
Brief Title: Once-weekly Petrelintide Versus Placebo for Obesity or Overweight With Co-morbidities
Acronym: ZUPREME
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP8396-23094; 2024-512549-18 (EudraCT Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: Weight management; Amylin analog
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Petrelintide Dose 1 (Experimental): Participants will self-inject petrelintide dose 1 subcutaneously once a week.
  Interventions: Drug: Petrelintide
- Petrelintide Dose 2 (Experimental): Participants will self-inject petrelintide dose 2 subcutaneously once a week.
  Interventions: Drug: Petrelintide
- Petrelintide Dose 3 (Experimental): Participants will self-inject petrelintide dose 3 subcutaneously once a week.
  Interventions: Drug: Petrelintide
- Petrelintide Dose 4 (Experimental): Participants will self-inject petrelintide dose 4 subcutaneously once a week.
  Interventions: Drug: Petrelintide
- Petrelintide Dose 5 (Experimental): Participants will self-inject petrelintide dose 5 subcutaneously once a week.
  Interventions: Drug: Petrelintide
- Placebo (Placebo Comparator): Participants will self-inject matching placebo to petrelintide subcutaneously once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Petrelintide — Petrelintide will be taken by participants once weekly as a self-administered subcutaneous injection.
  Other Names: ZP8396
  Arms: Petrelintide Dose 1; Petrelintide Dose 2; Petrelintide Dose 3; Petrelintide Dose 4; Petrelintide Dose 5
Drug: Placebo — Matching placebo to petrelintide will be taken by participants once weekly as a self-administered subcutaneous injection.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to compare dose levels of petrelintide versus placebo with regards to effect on body weight, safety, and tolerability.

DETAILED DESCRIPTION:
Obesity is a chronic disease with a rapidly increasing prevalence associated with significant comorbidities. Petrelintide is a long-acting amylin analog in development for weight management.

This is a randomized, double-blind, placebo-controlled, parallel-group, multinational, multicenter, dose-finding, Phase 2 clinical trial. The trial will compare 5 doses of once-weekly (OW) subcutaneously administered petrelintide with placebo.

This study consists of 3 periods:

1. A screening period of 2-3 weeks
2. A treatment period of 42 weeks
3. A safety follow-up period of 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants having body mass index (BMI) ≥30.0 kg/m2 or BMI ≥27.0 kg/m2 with the presence of at least one of the following comorbidities: hypertension or dyslipidemia (treated or untreated).
* A female participant is eligible to participate if she is:

  * A woman of nonchildbearing potential. OR
  * A woman of childbearing potential (WOCBP) who is not pregnant, does not intend to be pregnant, not lactating and is willing to use highly effective contraceptive methods (as required by local regulation or practice) throughout the trial and for 10 weeks after the last injection of the investigational medicinal product (IMP).
* Ability to comply with the protocol requirements including self-administration of IMP with vial and syringe.

Exclusion Criteria:

* Glycated hemoglobin (HbA1c) ≥48 mmol/mol (6.5%), as measured at screening.
* History of type 1 or type 2 diabetes mellitus.
* Treatment with glucose lowering agent(s) within 90 days prior to screening.
* A self-reported change in body weight >5% within 90 days prior to screening.
* Treatment with any medication (prescribed or over-the-counter) or alternative remedies (herbal or nutritional supplements) intended to promote weight loss within 6 months prior to screening.
* Previous or planned (during the trial period) obesity treatment with surgery or a body weight loss device. However, liposuction or surgical removal of fat depots more than 1 year prior to screening or device-based interventions (e.g. sleeve, banding or similar) that have been removed more than 6 months prior to screening, are allowed.
* Uncontrolled thyroid disease defined as thyroid stimulating hormone >4.20 mIU/L or <0.27 mIU/L as measured by the central laboratory at screening.
* Lifetime history of a suicidal attempt.
* History of major depressive disorder or other severe psychiatric disorders (e.g. schizophrenia or bipolar disorder).
* Estimated glomerular filtration rate value <60.0 mL/min/1.73m2, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) Creatinine Equation17, measured at screening.
* Impaired liver function, defined as alanine aminotransferase and/or aspartate aminotransferase ≥2.0 times or bilirubin >1.5 times upper normal limit, measured at screening.
* Presence or history of acute or chronic pancreatitis.
* Known clinically significant gastric emptying abnormality (for example, severe gastroparesis or gastric outlet obstruction) or chronic treatment that affects gastrointestinal (GI) motility.
* Presence or history of cardiovascular disease including stable and unstable angina pectoris, myocardial infarction, transient ischemic attack, stroke, cardiac decompensation.
* Presence or history of clinically significant arrhythmias or clinically significant conduction disorders.
* Known or suspected hypersensitivity to amylin analogs or related products.
* History of malignant neoplasms (except for basal or squamous cell skin cancer) within 5 years prior to screening.
* Known or suspected abuse of alcohol or recreational drugs.
* Participant previously treated with petrelintide or any other amylin analog.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in body weight to Week 28 | From Baseline (Day 1) to Week 28
  To compare the dose-response of increasing doses of petrelintide versus placebo on body weight, when added as an adjunct to a reduced-calorie diet and increased physical activity after 28 weeks of exposure.

SECONDARY OUTCOMES:
Percentage of Participants achieving ≥5% Body Weight Loss at Weeks 28 and 42 | From Baseline (Day 1) to Weeks 28 and 42
  To compare the efficacy of petrelintide versus placebo on body weight, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Percentage of Participants achieving ≥10% Body Weight Loss at Weeks 28 and 42 | From Baseline (Day 1) to Weeks 28 and 42
  To compare the efficacy of petrelintide versus placebo on body weight, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in body weight to Weeks 28 and 42 | From Baseline (Day 1) to Weeks 28 and 42
  To compare the efficacy of petrelintide versus placebo on body weight, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in waist circumference to Weeks 28 and 42 | From Baseline (Day 1) to Weeks 28 and 42
  To compare the efficacy of petrelintide versus placebo on waist circumference, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Percent change from baseline in body weight to Week 42 | From Baseline (Day 1) to Week 42
  To compare the efficacy of petrelintide versus placebo on body weight, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in hemoglobin A1c (HbA1c) to Week 42 | From Baseline (Day 1) to Week 42
  To compare the efficacy of petrelintide versus placebo on HbA1c, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in fasting glucose to Week 42 | From Baseline (Day 1) to Week 42
  To compare the efficacy of petrelintide versus placebo on fasting glucose, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in high-sensitivity C-reactive protein (hsCRP) to Week 42 | From Baseline (Day 1) to Week 42
  To compare the efficacy of petrelintide versus placebo on hsCRP, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Change from baseline in fasting lipids to Week 42 | From Baseline (Day 1) to Week 42
  To compare the efficacy of petrelintide versus placebo on fasting lipids, when added as an adjunct to a reduced-calorie diet and increased physical activity.
Number of treatment emergent adverse events (TEAEs) | From Baseline (Day 1) to Week 51
  To compare the safety and tolerability of petrelintide versus placebo when added as an adjunct to a reduced-calorie diet and increased physical activity.
Occurrences of anti-drug antibodies (ADAs) to petrelintide | From Baseline (Day 1) to Week 51
  To compare the safety and tolerability of petrelintide versus placebo when added as an adjunct to a reduced-calorie diet and increased physical activity.

CONTACTS AND LOCATIONS:
Locations (32):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Century Research LLC, Miami, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Great Lakes Clinical Trials LLC dba Flourish Research, Chicago, Illinois
  - AMR Wichita East, Wichita, Kansas
  - Alliance For Multispecialty Research, LLC, Lexington, Kentucky
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - CHEAR Center LLC, The Bronx, New York
  - Javara Inc, Charlotte, North Carolina
  - PharmQuest Life Sciences, LLC, Greensboro, North Carolina
  - Lucas Research, Inc., New Bern, North Carolina
  - AMR Norman, Norman, Oklahoma
  - Altoona Center for Clinical Research - Research, Duncansville, Pennsylvania
  - Alliance for Multispecialty Research, Knoxville, Tennessee
  - Clinical Trials of Texas, LLC., dba Flourish Research, San Antonio, Texas
  - Manaasas Clinical Research Center, Manassas, Virginia
- Poland (7):
  - Krakowskie Centrum MedyczneSp.z o.o, Krakow, Lesser Poland Voivodeship
  - ETG Siedlce, Siedlce, Masovian Voivodeship
  - FutureMeds Warszawa Centrum, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw, Masovian Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - FutureMeds Targowek, Warsaw, Masovian Voivodeship
  - Futuremeds Olsztyn, Olsztyn, Warmian-Masurian Voivodeship
- Romania (6):
  - Institutul National de Endocrinologie C I Parhon, Bucharest, București
  - Institutul Clinic Fundeni, Bucharest, București
  - Fundatia Dr Victor Babes, Bucharest, București
  - Institutul De Pneumoftiziologie Marius Nasta, Bucharest, București
  - Spitalul Clinic Judetean de Urgenta Sf Apostol Andrei Constanta, Constanța, Constanța County
  - Top Diabet, Craiova, Dolj

IPD SHARING:
Plan to Share IPD: No